CLINICAL TRIAL: NCT01109576
Title: Pilot Study: Self Management Groups for Veterans With Dual Sensory Loss
Brief Title: Workshops for Veterans With Vision and Hearing Loss
Acronym: DSLW
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C7460-P
Record Dates: First submitted 2010-04-19; First posted 2010-04-23 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-08

CONDITIONS: Deafness; Blindness
Keywords: deafness-blindness; pilot study; self management education; dual sensory loss; rehabilitation; peer support groups; age related
MeSH Terms: conditions — Deafness; Blindness; Deaf-Blind Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSL workshop participants (Experimental): Three to five Veterans with DSL.
  Interventions: Behavioral: DSL Workshop

INTERVENTIONS:
Behavioral: DSL Workshop — A series of 6 weekly 2 hour interactive workshops for Veterans with age-related Dual Sensory Loss that provide instruction, skills training, exercises and facilitated interaction among peers.
  Other Names: Dual Sensory Loss Self Management Groups

SUMMARY:
This is a pilot study of workshops to help Veterans with both vision and hearing loss live a happier, fuller and less stressful life. The results will be used to guide the development of a large scale clinical trial.

DETAILED DESCRIPTION:
This pilot study will enrolled 13 Veterans with Dual Sensory Loss (DSL), age 65 to over 89. The project headquarters in the Portland Oregon Veterans Affairs Medical Center will be tasked with the development of the workshops and writing of a Curriculum and Procedures Manual. The Atlanta VAMC research collaborators enrolled the 13 Veterans. Staff turnover reduced time available for enrollment and data collection. We therefore eliminated the original comparison group design and this study had only one experimental intervention arm and no control intervention or other arm. Veterans were chronologically enrolled who responded to recruitment letters and who passed telephone and onsite screening. The intervention consisted of six weekly two hour workshops providing information, skills training and exercises about self-managing DSL effects on daily life. Preliminary effectiveness data was collected and analyzed, and a large scale clinical trial will be proposed as a followup to explore the efficacy of this management approach. This study data tracked pre and post intervention within subject changes.

ELIGIBILITY:
Inclusion Criteria:

* Veteran;
* Vision loss > 20/70 better eye;
* Hearing loss > 40 decibels better ear;
* Cognition Within Normal Limits (WNL);
* No behavioral flag or psychiatric diagnosis;
* Documented psychosocial restrictions secondary to vision and hearing loss

Exclusion Criteria:

* Vision and/or hearing can be corrected by surgical or pharmacological treatment;
* Requires use of sign language interpreter

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel Turbin, PhD, Principal Investigator — Veterans Health Administration (VHA)
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - VA Portland Health Care System, Portland, OR, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- DSL Workshop Participants: Three to five Veterans with DSL.
  DSL Workshop: A series of 6 weekly 2 hour interactive workshops for Veterans with age-related Dual Sensory Loss that provide instruction, skills training, exercises and facilitated interaction among peers.
  Participant Flow Completed: Twelve participants completed the entire protocol, including all outcomes measures.
Period: Overall Study
Arm/Group | DSL Workshop Participants
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | DSL Workshop Participants
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 85 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 13
Profiles of Mood States Total Score [Mean (Standard Deviation); unit: units on a scale] — The Profile of Mood States contains 65 self-reported items in 6 subscales (Tension, Depression, Anger, Vigor, Fatigue, and Confusion). Items are rated using a 5-point Likert Scale (scale: 0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely). Total mood disturbance is calculated by subtracting the Vigor subscale score from the sum of the Tension, Depression, Anger, Fatigue, and Confusion subscale scores. Total scores can range from -32 to 200, with higher score indicating more mood disturbance.
  units on a scale | 16 (26.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Profile of Mood States Total Score.
Description: The change in Profile of Mood States total score is defined as the 8 week follow-up total score minus the baseline POMS total score. The scale measures change in mood states before and after treatment. The change score can range from -232 to 232, with negative values indicating greater reduction in emotional distress.
Time Frame: Change in Profile of Mood States Score from Baseline to 8 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DSL Workshop Participants
Number analyzed (Participants) | 12
units on a scale | 4.5 (21.9)

ADVERSE EVENTS:
Groups:
- DSL Workshop Participants: Dual Sensory Loss (DSL) workshop participants. Three to five Veterans with DSL.
  DSL Workshop: A series of 6 weekly 2 hour interactive workshops for Veterans with age-related Dual Sensory Loss that provide instruction, skills training, exercises and facilitated interaction among peers.
Arm/Group | DSL Workshop Participants
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DSL Workshop Participants (N=13)
suicidal ideations (Psychiatric disorders) | 1 (1) — One veteran participant presented with clinically significant depression and verbalized suicidal ideation to the study coordinator and subsequently was referred to the Suicide Prevention Coordinator at the Atlanta Veterans Affairs Medical Center.

LIMITATIONS AND CAVEATS:
The sample size was too small to draw any definitive conclusion from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes